CLINICAL TRIAL: NCT06623942
Title: Prostasin Levels in Preeclampsia: A Comparative Study With Healthy Pregnancies
Brief Title: Prostasin Levels in Preeclamptic Women
Status: Completed | Type: Observational
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Principal Investigator, Gökhan Bolluk, MD, Başakşehir Çam & Sakura City Hospital
Other Study IDs: ProstasinStudy
Record Dates: First submitted 2024-09-24; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Pre-Eclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 (Control): This group consists of uncomplicated pregnancies (who do not have pre-eclampsia or severe pre-eclampsia). These participants will be matched to the case group based on relevant characteristics such as age, gestational age, and other demographic factors.
- Group 2 (Case - Pre-eclampsia): This group consists of pregnant women diagnosed with pre-eclampsia and severe preeclampsia.

SUMMARY:
This study will aim to compare maternal serum prostasin levels between women diagnosed with preeclampsia and healthy normotensive pregnant controls. Participants will be divided into two main groups: those with preeclampsia and those with uncomplicated pregnancies. The preeclampsia group will further be subdivided based on the severity of the condition. Maternal serum samples will be collected from all participants, and prostasin levels will be measured using ELISA. Statistical analyses will be performed to evaluate whether prostasin levels are significantly elevated in the preeclampsia group, particularly in those with severe features, and to assess its potential as a biomarker for the condition.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Preeclampsia: Defined by new-onset hypertension (systolic Blood Pressure ≥140 mmHg and/or diastolic Blood Pressure ≥90 mmHg) after 20 weeks of gestation, with or without proteinuria.
* Control Group: Healthy pregnancies without preeclampsia or other significant maternal or fetal complications.

Exclusion Criteria:

* Multiple Pregnancies
* Pregestational Diabetes
* Chronic Hypertension
* Systemic Diseases (Chronic kidney disease, autoimmune diseases)
* Fetal Anomalies
* Premature Rupture of Membranes.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The groups in this study will be selected consists of pregnant women receiving care at a referral center for maternal care.
Sampling Method: Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Maternal Serum Prostasin Levels | Up to 8 weeks (Patients will be followed from inclusion in the study until the end of their pregnancy.
  To compare Prostasin Levels between the pre-eclampsia and the control group.

CONTACTS AND LOCATIONS:
Locations (1):
- Cam and Sakura City Hospital, Istanbul, Turkey (Türkiye)